CLINICAL TRIAL: NCT00760409
Title: Prospective Study Differentiating Recurrent Brain Tumor Versus Radiation Injury Using Magnetic Resonance (MR) Spectroscopy, Diffusion Tensor Imaging and Diffusion Weighted Imaging on 3T(Tesla) MR Scanner
Brief Title: Differentiating Recurrent Brain Tumor Versus Radiation Injury Using MRI
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Pia C Maly Sundgren, MD, PhD, Principal Investigator, University of Michigan
Other Study IDs: HUM00050584
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Radiation Injury; Brain Tumor
Keywords: recurrent tumor
MeSH Terms: conditions — Radiation Injuries; Brain Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Radiation Injury: Radiation Injury Recurrent symptoms after radiation therapy of a brain tumor are not always the result of tumor recurrence but may represent radiation necrosis of the brain.
- Tumor Recurrence: Symptoms are the result of actual tumor recurrence

SUMMARY:
The purpose of this study is to determine if certain MRI imaging sequences (pictures) are more helpful to the physicians in determining if a brain tumor has recurred or if the person has radiation injury following their treatment.

DETAILED DESCRIPTION:
After a patient has been treated for a brain tumor by radiation the area of the brain that has been treated changes in appearance. These changes in appearance can make it hard to determine if a brain tumor has come back at the same site or if it is radiation injury. The purpose of this study is to determine if certain MRI imaging sequences (pictures) are more helpful to the physicians in determining if the tumor has come back or if it is radiation injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously treated with radiation therapy (including radiosurgery), with or without previous surgery or chemotherapy, with a new contrast enhancing lesion(s) with the size of 1 cm or more on conventional brain MRI examination are eligible
* Patients must have a previously histological confirmed brain tumor
* Patients must be 18 years of age or older
* Patients must sign a study-specific consent form approved by the Institutional Review Board of the University of Michigan indicating prior to study entry

Exclusion Criteria:

* Pregnant woman
* For the purpose of this radiological study and in collecting data from the patient but not from receiving the MR Spectroscopy if it is clinically indicated.
* Patients unable to undergo MRI imaging because of non-compatible devices such as cardiac pacemakers, other implanted electronic devices, or foreign body in the eye
* Also patients with metallic prostheses, or ferromagnetic prostheses (e.g. pins in artificial joints and surgical pins/clips in the face or skull region), or patients with braces since these devices may cause metal artifacts which may obscure the images and result in artifacts on the MR spectroscopy.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have had a previous brain tumor and their physician has ordered a follow up MRI because your tumor may have returned.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-09; Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging of treated brain tumors | 6mth. and 1 year follow-up
  The purpose of this study is to determine if certain MRI imaging sequences are more helpful to the physicians in determining if the tumor has come back or if it is radiation injury

CONTACTS AND LOCATIONS:
Overall Officials: Pia M Sundgren, MD, Ph.D, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No